CLINICAL TRIAL: NCT06988306
Title: Randomized Controlled Trial of Lifestyle Interventions for the Prevention of Diabetes in US Home Visiting Programs
Brief Title: Lifestyle Interventions to Prevent Diabetes in U.S. Home Visiting Programs
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: California Polytechnic State University-San Luis Obispo (Other)
Collaborators: Lifespan/ The Miriam Hospital (Unknown); Northwestern University (Other); Bradley Hospital (Other); Patient-Centered Outcomes Research Institute (Other)
Responsible Party: Principal Investigator, Suzanne Phelan, Professor, California Polytechnic State University-San Luis Obispo
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 2025-056; MMM-2024C1-37760 (Other Grant/Funding Number: Patient-Centered Outcomes Research Institute)
Record Dates: First submitted 2025-04-06; First posted 2025-05-23 (Actual); Last update posted 2025-07-14 (Actual); Status verified 2025-07

CONDITIONS: Diabetes Mellitus; Gestational Diabetes Mellitus (GDM)
Keywords: medically tailored meals; gestational diabetes; food is medicine; home visiting
MeSH Terms: conditions — Diabetes Mellitus; Diabetes, Gestational | interventions — Meals

STUDY DESIGN:
Who Masked: Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Usual Home Visiting plus GDM Enhanced (Active Comparator): This group receives usual home visitation plus GDM Enhanced intervention.
  Interventions: Behavioral: GDM Enhanced
- Usual HV + GDM Enhanced + Meals (Experimental): This group will receive usual home visitation plus GDM Enhanced plus medically tailored meals.
  Interventions: Behavioral: GDM Enhanced; Behavioral: Meals

INTERVENTIONS:
Behavioral: GDM Enhanced — The GDM Enhanced intervention is comprised of HV-delivered, evidence-based modules (10-20 minutes) with facilitator guides. The content prioritizes management and prevention of diabetes through healthy eating, physical activity, and stigma-informed weight management strategies.
Behavioral: Meals — The Meal intervention includes medically tailored meals being provided to participants starting after randomization and tailored to their individual dietary preferences and cultural considerations.
  Arms: Usual HV + GDM Enhanced + Meals

SUMMARY:
The study is examining the health effects of gestational diabetes mellitus (GDM) intervention and medically tailored meals within home visiting. A large study is proposed that will include nearly a thousand pregnant or recently pregnant adults with recent GDM and who are from different regions and backgrounds. Two treatment approaches are compared, and both are in home visiting. One treatment group is receiving enhanced lifestyle support for GDM along with meals, and the other is receiving just the enhanced lifestyle support. The study will examine whether these interventions help reduce diabetes and pre-diabetes through 12 months postpartum, as well as other health factors like weight and blood pressure.

DETAILED DESCRIPTION:
Gestational diabetes mellitus (GDM) is rapidly rising in prevalence and has been linked with several short and long-term adverse maternal health outcomes, including type 2 diabetes (T2DM) and cardiovascular disease. The postpartum year is a time of heightened risk, and 32-46% of people with GDM develop type 2 diabetes (T2DM) or Pre-Diabetes (PreDM) during the postpartum year. To prevent maternal diabetes, US guidelines recommend behavioral counseling to promote healthy eating, activity, and weight, but dissemination channels have been lacking. Evidence-based home visiting programs, with their well-established infrastructure in every state and focus on maternal and child health, are a promising platform through which the recommended behavioral interventions could reach people with GDM and reduce health disparities. Effective GDM intervention within home visiting needs to be potent, build on existing content, and remain brief, so as not to displace other evidence-based content. Integrating referral to medically tailored meals (MtMs) is a Food is Medicine strategy that may prevent and mitigate maternal diabetes in home visiting. Access to MtMs has been expanding rapidly in the US, with 10 states currently having and 5 states pending Medicaid Service waivers that offer coverage for MtMs. Systematic reviews have found that providing MtMs allows patients to experience significantly better glucose and weight management, improved food insecurity and dietary quality, and greater treatment satisfaction. MtMs also benefit health systems, insurers, and governments through reduced costs and fewer hospitalizations and emergency department visits. However, national calls and systematic reviews have identified a major evidence gap and the need for adequately powered effectiveness trials to determine whether MtMs are effective in treating and preventing maternal diabetes. For MtMs to continue as a treatment approach for GDM, compelling evidence is needed that they work and for whom and in what context. The primary aim of this study is to evaluate the 12-month incidence T2DM/PreDM in people with GDM who receive GDM Enhanced + Meals vs. GDM Enhanced Only within home visiting. A robust implementation process evaluation will inform ensure successful sustainment and reach for diverse pregnant and postpartum people with GDM. A Hybrid Type 1 effectiveness-implementation trial is proposed. The study will recruit 978 perinatal, English or Spanish-speaking adults nationwide from three clinical centers serving the West, Midwest/South, and East regions. Home visiting clients (35% Black; 40% Hispanic) with recent GDM diagnosis and will be randomized within site and home visiting agency to one of two treatment arms: GDM enhanced lifestyle intervention plus MtMs (GDM Enhanced + Meals) or GDM Enhanced Only. The primary study aim is to evaluate the 12-month incidence of T2DM/PreDM. Secondary aims will examine treatment group differences in health factors (weight, blood pressure) and client-centered outcomes (diet quality, physical activity, home food environment, food security, quality of life, treatment satisfaction, self-efficacy, mood) at 3, 6, and 12 months postpartum. Key moderators (Black/White race, Hispanic/Non-Hispanic ethnicity, food security), and mediators (changes in weight, dietary quality, physical activity, and the home food environment) will be identified. The RE-AIM framework will guide an implementation process evaluation to plan for successful delivery and sustainment of the interventions. Findings from this from large scale, adequately powered trial of MtMs for maternal health will fill a major gap in the literature. If the MTM approach is found effective, there will be strong justification to bolster access (at state level) and referrals (within home visiting) to MtMs. Findings will inform tailored strategies to ensure successful sustainment in home visiting and reach for diverse pregnant and postpartum people with GDM.

ELIGIBILITY:
Inclusion Criteria:

* Currently in home visiting
* Pregnant or < 3 months (13 weeks) postpartum
* Gestational Diabetes Mellitus diagnosis in most recent pregnancy (based on self-report)
* Aged 18 years or older
* English- or Spanish-speaking.
* Not currently being given medically tailored meals
* Willing to receive randomization to either group

Exclusion Criteria:

• Pre-existing diabetes (based on self-report)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 978 (Estimated)
Dates: Start 2026-01-31 (Estimated); Primary Completion 2030-04-30 (Estimated); Study Completion 2030-04-30 (Estimated)

PRIMARY OUTCOMES:
Diabetes/Pre-Diabetes | From enrollment to 12 months postpartum
  The Primary Outcome Measure in this study is a categorical outcome of glucose tolerance (i.e., healthy glucose tolerance vs. type 2 diabetes/pre-diabetes) at 12 months postpartum. The test will be conducted at CLIA-certified lab. A 2-hour oral glucose tolerance test (OGTT) will characterize people into one of two categories: 1) healthy glucose tolerance; or 2) type 2 diabetes (2-hour post 75g load glucose level of 200 mg/dL or greater) or pre-diabetes (a 2-hour post 75g load glucose level of 140 to 199 mg/d).

SECONDARY OUTCOMES:
HbA1c concentration | From enrollment to 3, 6, and 12 months postpartum
  HbA1c will be measured utilizing an at-home test kit (finger-stick, whole-blood test)
Systolic blood pressure | From enrollment to 3, 6, and 12 months postpartum
  Systolic blood pressure will be self-measured in the home with trained research assistants guiding the assessment
Diastolic blood pressure | From enrollment to 3, 6, and 12 months postpartum
  Diastolic blood pressure will be self-measured in the home with trained research assistants guiding the assessment
Body weight | From enrollment to 3, 6, and 12 months postpartum
  Body weight is obtained using remote scales provided to participants.
Child zBMI | From 3 months to 6 and 12 months
  Remote, guided parent measurements of child weight and length will be used to calculate the child's body mass index z-score (zBMI), along with parent-reported infant sex.
Diet quality | From enrollment to 3, 6, and 12 months postpartum
  The Automated Self-Administered (ASA) 24-hour Recall of the National Cancer Institute will be used by trained staff to obtain an interview-based assessment of dietary quality. Healthy Eating Index (HEI) scores will be calculated by linking ASA24 output to the HEI scoring algorithm, which evaluates diet quality based on alignment with the Dietary Guidelines for Americans.Scores range from 0 to 100.
Metabolic equivalent task minutes per week of moderate-to-vigorous physical activity | From enrollment to 3, 6, and 12 months postpartum
  The International Physical Activity Questionnaire will be used to measure metabolic equivalent task (MET)-minutes per week of moderate-to-vigorous physical activity. Scores range from 0 to >10,000 MET-minutes/week, with higher scores indicating greater physical activity, which is considered a better outcome.
Home Food Environment | From enrollment to 3, 6, and 12 months postpartum
  The home food environment checklist will be used to measure number of healthy foods in the home. Higher scores indicate a greater number of healthy foods present.
Food Security | From enrollment to 3, 6, and 12 months postpartum
  The U.S. Household food security survey will be used to measure a categorical classification or high food security, marginal food security, low food security, and very low food security
Global Physical Health | From enrollment to 3, 6, and 12 months postpartum
  The Patient-Reported Outcomes Measurement Information System (PROMIS) Global Health 10-item scale will be used to assess Global Physical Health (GPH). Raw scores are converted to T-scores, standardized to the U.S. general population (mean = 50, SD = 10). T-scores typically range from 20 to 80, with higher scores indicating better health.
Global Mental Health | From enrollment to 3, 6, and 12 months postpartum
  The Patient-Reported Outcomes Measurement Information System Global Health 10-item scale will be used to assess Global Mental Health. Raw scores are converted to T-scores, standardized to the U.S. general population (mean = 50, SD = 10). T-scores typically range from 20 to 80, with higher scores indicating better health.
Nutrition Self-Efficacy | From enrollment to 3, 6, and 12 months postpartum
  The Nutrition Self-Efficacy Scale will be used to assess participants' confidence in their ability to engage in healthy eating, yielding a continuous self-efficacy score. Each item is rated on a 5-point Likert scale from 1 (not at all confident) to 5 (very confident), resulting in a total score range of 10 to 50. Higher scores reflect greater self-efficacy for healthy eating behaviors
Center for Epidemiologic Studies Depression Scale | From enrollment to 3, 6, and 12 months postpartum
  The Center for Epidemiologic Studies Depression Scale - 10-item version (CES-D-10) will be used to assess depressive symptoms. Each item is rated on a 4-point Likert scale from 0 (rarely or none of the time) to 3 (most or all of the time), yielding a total score range of 0 to 30. Higher scores indicate greater depressive symptomatology.
Barriers to Healthy Eating | From enrollment to 3, 6, and 12 months postpartum
  Barriers to Healthy Eating Questionnaire is 14-items and assesses perceived barriers to healthy eating. The total score is calculated by summing all 14 items. Total scores range from 0 to 14, with higher scores reflecting greater overall perceived barriers to following a healthy eating pattern.

OTHER OUTCOMES:
Feasibility of Intervention Measure | 12 months postpartum
  The Feasibility of Intervention Measure will be used to assess participants' perceptions of how feasible the intervention is to implement. The scale includes 4 items, each rated on a 5-point Likert scale from 1 (completely disagree) to 5 (completely agree), resulting in a total score range of 4 to 20. Higher scores indicate greater perceived feasibility of the intervention.
Acceptability of Intervention Measure | 12 months postpartum
  The Acceptability of Intervention Measure (AIM) will be used to assess participants' perceptions of how acceptable the intervention is. The measure includes 4 items, each rated on a 5-point Likert scale from 1 (completely disagree) to 5 (completely agree), resulting in a total score range of 4 to 20. Higher scores indicate greater acceptability of the intervention.
Intervention Appropriateness Measure | 12 months postpartum
  The Intervention Appropriateness Measure (IAM) will be used to assess participants' perceptions of how suitable the intervention is. The scale consists of 4 items, each rated on a 5-point Likert scale from 1 (completely disagree) to 5 (completely agree), yielding a total score range of 4 to 20. Higher scores indicate greater perceived appropriateness of the intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Suzanne Phelan, PhD, Principal Investigator — California Polytechnic State University-San Luis Obispo
Locations (3):
- United States (3):
  - California Polytechnic State University, San Luis Obispo, California
  - Northwestern University, Chicago, Illinois
  - Miriam Hospital, Providence, Rhode Island

IPD SHARING:
Plan to Share IPD: Yes
We will share de-identified individual participant data related to primary and secondary outcomes. These data may include measures of diabetes, physical activity, diet quality, and other health indicators.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: April, 2031
Access Criteria: Data will be made available to qualified researchers upon reasonable request and completion of a data use agreement that protects participant confidentiality and outlines permitted uses of the data.